CLINICAL TRIAL: NCT06508619
Title: Blood Pressure Treatment by the Corsano CardioWatch 287-2 Evaluation Study
Acronym: BPTreat
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Corsano Health B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: BPTreat
Record Dates: First submitted 2024-06-07; First posted 2024-07-18 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2024-07

CONDITIONS: High Blood Pressure
Keywords: Remote monitoring; Photoplethysmography; Blood pressure; Blood pressure lowering medication; Wearable technology; Evaluation
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients receiving blood pressure lowering medication (uptitration) as standard of care (Experimental): Patients receiving blood pressure lowering medication (uptitration) as standard of care
  Interventions: Device: Corsano CardioWatch 287-2 non-invasive blood pressure (NIBP) monitoring

INTERVENTIONS:
Device: Corsano CardioWatch 287-2 non-invasive blood pressure (NIBP) monitoring — Patients receive Corsano CardioWatch 287-2 for continous NIBP monitoring and perform several spot-checks using an automated BP cuff as a reference during the start or uptitration of BP lowering medication

SUMMARY:
Rationale: Wearables have the potential to monitor patients remotely. The Corsano CardioWatch 287-2 is such a medical device that can monitor long-term blood pressure. The device has been validated using clinical trials in hospitals, but evaluation in the intended remote setting during treatment is lacking.

Primary objective: To assess the ability to track blood pressure decrease measured by the Corsano CardioWatch 287-2 after a period of 28 days of antihypertensive drug treatment initiation, uptitration or change in antihypertensive drugs.

Study population: A group, untreated or treated for hypertension, with uncontrolled BP and medical indication for antihypertensive drug treatment initiation, uptitration or change in antihypertensive drugs.

Study design: Blood pressure will be measured by the investigative device and a reference device at pre-treatment and after 28 days. The investigative device is the Corsano CardioWatch 287-2, which measures blood pressure through optical photoplethysmography (PPG). The reference method involves automatic blood pressure cuff measurements.

Main study parameters/endpoints: Absolute systolic and diastolic blood pressure decrease after change of treatment measured by the Corsano Cardiowatch 287-2 after 28 days, compared to automatic blood pressure cuff measurements.

DETAILED DESCRIPTION:
Background and Introduction:

Blood pressure (BP) is a cardiovascular risk factor that affects millions of people worldwide. BP is a major determinant of stroke, heart failure, coronary artery disease, and chronic kidney disease [1]. Hypertension may be asymptomatic or episodic. Accurate monitoring of BP is required to tailor medication to the patient's specific needs to maintain blood pressure control [2]. Therefore, accurate and continuous monitoring of BP is crucial for optimal diagnosis, treatment, and prevention of cardiovascular events.

However, conventional methods for measuring BP have several limitations. Most BP monitors use an occluding cuff that inflates periodically to obtain intermittent readings. Cuff measurements may not reflect the true BP variations that occur throughout the day and night due to various factors such as physical activity, stress level or sleep quality [3].

Wearable devices are emerging as a promising alternative to conventional methods for measuring BP [4, 5, 6]. They can measure BP continuously and non-invasively by using novel sensors and algorithms that do not require a cuff or electrodes. Wearable devices can also enable remote monitoring and data transmission to healthcare providers or researchers. However, wearable devices need to be evaluated against standard methods in different clinical settings and patient populations.

The Corsano CardioWatch 287-1 conforms with the European Medical Device Regulation (CE-MDR) and is a clinically validated vital signs monitoring bracelet. It is able to continuously measure pulse rate [6], inter-beat intervals [6], breathing rate [7], sleep and activity. The Corsano CardioWatch 287-2, an iteration on the 287-1, adds electrocardiogram (ECG), oxygen saturation (SpO2), galvanic skin response (GSR), core body temperature and non-invasive blood pressure (NIBP).

The Corsano CardioWatch Corsano 287-2 has been submitted to laboratory tests against internationally recognized standards for the monitoring of pulse rate, respiratory rate, SpO2, GSR, temperature and ECG. Additionally, the MULTI-VITAL study (NL80236.000.22) has clinically validated Corsano 287-2 in a controlled intramural healthcare setting. The Remote Cardiac Monitoring (RECAMO) study is underway to assess the free-living remote care setting long-term monitoring validity using a static test. Clinical evaluation in a non-static remote care setting is still lacking, however.

Antihypertensive drugs reduce BP through blood volume reduction and vasodilatation which are very different physiological mechanisms. This consequently changes the PPG waveform in distinct ways which constitutes a necessarily challenging test for cuffless devices. The accuracy of the Corsano CardioWatch 287-2 during a change of antihypertensive treatment has not yet been evaluated. However it is an important target for future use of the CardioWatch 287-2. Additionally, it is a recommended research in the European Society of Hypertension (ESH) recommendations for the validation of cuffless blood pressure measuring devices [8].

The current trial aims to clinically assess the Corsano CardioWatch 287-2 on blood pressure monitoring during antihypertensive treatment in a remote care setting.

Objectives:

The main objective is to assess the Corsano CardioWatch 287-2's ability to track blood pressure decrease over a period of 28 days after antihypertensive drug treatment initiation, uptitration or change in antihypertensive drug.

The assessment is done by comparing the blood pressure measurements of the Corsano CardioWatch 287-2 with those of an automatic cuff.

Study Design:

Patients who are untreated or treated for hypertension, with uncontrolled BP and medical indication for antihypertensive drug treatment initiation, uptitration, or change in antihypertensive drugs will be approached for participation in the trial. The ability of the CardioWatch 287-2 to track decreases in blood pressure will be assessed. Blood pressure measured by the CardioWatch 287-2 at the beginning and end of the study period will be compared with the blood pressure measured by a reference device, which is an automatic blood pressure cuff. Blood pressure will be measured continuously by the Corsano CardioWatch 287-2 during 28 days. These measurements are only meant for study purposes and not part of standard care.

Blood pressure measurements with the Corsano cuff (an automatic oscillometric blood pressure monitoring device) will be used for initialization of the Corsano CardioWatch 287-2 on day 0. On day 1, the antihypertensive drug treatment initiation, uptitration, or change in antihypertensive drug will be started. The automatic blood pressure cuff measurements at day 0 and 28 will be used to assess the CardioWatch's accuracy by comparing it to the closest available blood pressure measurement by the CardioWatch.

The mean difference in blood pressure decrease between the Corsano CardioWatch 287-2 and reference automatic blood pressure cuff will be analyzed.

Study population:

The study will involve a patient group visiting the outpatient cardiology clinic at the Reinier de Graaf Gasthuis. This group has an uncontrolled BP and therefore medical indication for antihypertensive drug treatment initiation, uptitration, or change in antihypertensive drugs.

Sample size calculation:

The participants will be included with the aim to assess the long-term variation in blood pressure during antihypertensive treatment. Sample size calculation for the assessment of blood pressure monitoring is based on Association for the Advancement of Medical Instrumentation/European Society of Hypertension/International Organization for Standardization (AAMI/ESH/ISO) consensus that at least 35 patients are required for the validation of a 'moderate accuracy' device and recommends the following criteria to be met [8]:

* Males ≥ 30 % and females ≥ 30 %
* Subjects with an added diuretic drug ≥ 35%
* Subjects with an added long-acting dihydropyridine calcium channel blocker ≥ 35%
* ≥ 60% of the subjects need a reference systolic BP decrease ≥ 10 mmHg
* ≥ 60% of the subjects need a reference diastolic BP decrease ≥ 5 mmHg
* ≥ 30% of the subjects need a reference systolic BP decrease < 10 mmHg
* ≥ 30% of the subjects need a reference diastolic BP decrease < 5 mmHg Based on prior studies conducted by Corsano, e.g. RECAMO Study, the investigators experienced difficulty in obtaining a diverse study group in terms of inclusion requirements. To meet these criteria the investigators will include at least 80 patients.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 80 years old;
* able to provide consent;
* untreated or treated for hypertension, with uncontrolled BP and medical indication for antihypertensive drug initiation or uptitration or change in antihypertensive drug per doctor prescription.

Exclusion Criteria:

* Unable to wear the Corsano CardioWatch 287 due to reasons such as allergic reactions, wounds, amputations etc.;
* Unable to receive blood pressure measurements per cuff due to lymphedema, amputation, dialysis shunt, wounds, etc.;
* Pregnant women;
* Breastfeeding women;
* Upper arm circumference not within the cuff range (22-42 cm)
* Unable or not willing to sign for informed consent;
* Significant mental or cognitive impairment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-02 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Baseline average BP for both CardioWatch 287-2 and reference | Measured in each patient on 1st study day
  Baseline average blood pressure per patient and its standard deviation measured by automatic blood pressure cuff reference device and CardioWatch 287-2, separately.
Post-treatment average BP for both CardioWatch 287-2 and reference | Measured in each patient on 28th/last study day
  Post-treatment average blood pressure and its standard deviation measured by automatic blood pressure cuff reference device and CardioWatch 287-2, separately.
Average BP change comparing CardioWatch 287-2 and reference | Measured in each patient on 28th/last study day
  Absolute systolic and diastolic BP decrease and its standard deviation after change of treatment measured by the Corsano CardioWatch 287-2 after 28 days of monitoring, compared to automatic blood pressure cuff measurements.

SECONDARY OUTCOMES:
Bland-Altman for CardioWatch 287-2 vs. reference BP | Measured in each patient on 28th/last study day
  Mean bias and limits of agreement between blood pressure measurements measured by the Corsano CardioWatch 287-2 and blood pressure measured by an automatic blood pressure cuff using a Bland Altman analysis.
Pearson correlation coefficient between CardioWatch 287-2 vs. reference BP | Measured in each patient on 28th/last study day
  Pearson correlation coefficient between blood pressure decrease measured by the Corsano CardioWatch 287-2 and blood pressure decrease measured by an automatic blood pressure cuff.

CONTACTS AND LOCATIONS:
Overall Officials: Eelko Ronner, PhD, Principal Investigator — Reinier de Graaf Groep
Locations (1):
- Reinier de Graaf Gasthuis, Delft, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Michaud GF, Stevenson WG. Atrial Fibrillation. N Engl J Med. 2021 Jan 28;384(4):353-361. doi: 10.1056/NEJMcp2023658. No abstract available. PMID 33503344
- [Background] Sheppard JP, Lown M, Burt J, Ford GA, Hobbs FDR, Little P, Mant J, Payne RA, McManus RJ; OPTiMISE Investigators. Blood Pressure Changes Following Antihypertensive Medication Reduction, by Drug Class and Dose Chosen for Withdrawal: Exploratory Analysis of Data From the OPTiMISE Trial. Front Pharmacol. 2021 Apr 20;12:619088. doi: 10.3389/fphar.2021.619088. eCollection 2021. PMID 33959004
- [Background] Meidert AS, Saugel B. Techniques for Non-Invasive Monitoring of Arterial Blood Pressure. Front Med (Lausanne). 2018 Jan 8;4:231. doi: 10.3389/fmed.2017.00231. eCollection 2017. PMID 29359130
- [Background] Sessler DI, Saugel B. Beyond 'failure to rescue': the time has come for continuous ward monitoring. Br J Anaesth. 2019 Mar;122(3):304-306. doi: 10.1016/j.bja.2018.12.003. Epub 2019 Jan 3. No abstract available. PMID 30770047
- [Background] McGillion MH, Duceppe E, Allan K, Marcucci M, Yang S, Johnson AP, Ross-Howe S, Peter E, Scott T, Ouellette C, Henry S, Le Manach Y, Pare G, Downey B, Carroll SL, Mills J, Turner A, Clyne W, Dvirnik N, Mierdel S, Poole L, Nelson M, Harvey V, Good A, Pettit S, Sanchez K, Harsha P, Mohajer D, Ponnambalam S, Bhavnani S, Lamy A, Whitlock R, Devereaux PJ; PROTECT Network Investigators. Postoperative Remote Automated Monitoring: Need for and State of the Science. Can J Cardiol. 2018 Jul;34(7):850-862. doi: 10.1016/j.cjca.2018.04.021. Epub 2018 Apr 25. PMID 29960614
- [Background] Blok S, Piek MA, Tulevski II, Somsen GA, Winter MM. The accuracy of heartbeat detection using photoplethysmography technology in cardiac patients. J Electrocardiol. 2021 Jul-Aug;67:148-157. doi: 10.1016/j.jelectrocard.2021.06.009. Epub 2021 Jul 2. PMID 34256184
- [Background] Gehring JM, Saeijs-van Niel LC, Ten Bosch-Paniagua LP, Frank MH. Continuous respiration rate monitoring using photoplethysmography technology in patients with Obstructive Sleep Apnea. Under peer review
- [Background] Stergiou GS, Avolio AP, Palatini P, Kyriakoulis KG, Schutte AE, Mieke S, Kollias A, Parati G, Asmar R, Pantazis N, Stamoulopoulos A, Asayama K, Castiglioni P, De La Sierra A, Hahn JO, Kario K, McManus RJ, Myers M, Ohkubo T, Shroff SG, Tan I, Wang J, Zhang Y, Kreutz R, O'Brien E, Mukkamala R. European Society of Hypertension recommendations for the validation of cuffless blood pressure measuring devices: European Society of Hypertension Working Group on Blood Pressure Monitoring and Cardiovascular Variability. J Hypertens. 2023 Dec 1;41(12):2074-2087. doi: 10.1097/HJH.0000000000003483. Epub 2023 Jun 22. PMID 37303198